CLINICAL TRIAL: NCT05191030
Title: Food Insecurity, Poor Diet, and Metabolic Syndrome: Cortisol's Amplifying Role
Brief Title: Cortisol and Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, A. Janet Tomiyama, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-000048; R01DK128575 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Food Insecurity
Keywords: Food insecurity; Physiological Stress; Psychological Stress; Cortisol; Eating; Diet
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The study is a within-subjects experiment. The order in which participants undergo the experimental or control conditions/arms will be counterbalanced. 50% of participants will undergo the experimental condition first and then the control condition, one month later. The rest of the sample will undergo the control condition first then the experimental condition, one month later.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (High-Stress) Arm (Experimental): Participants undergoing the experimental (high-stress) arm are exposed to a gold-standard laboratory stressor, the Trier Social Stress Test (Kirschbaum et al., 1993). Participants are given five minutes to prepare for a five-minute speech task followed by a five-minute mental arithmetic task in front of two panelists wearing white lab coats (i.e., a male and female research assistant). The speech task posits the participant in a mock interview, with the two panelists listening to the speech in an unresponsive, neutral manner and asking standardized probing questions. Participants undergoing the mental arithmetic task are instructed to subtract odd numbers (i.e., 7 and 13) from a large number (i.e., 2935) as quickly as possible. If the participant makes a mistake, the panelist interrupts them and instructs them to start the task again from the beginning. The panelists also constantly remind the participant to "go faster" if they start to slow down with the task.
  Interventions: Behavioral: High-Stress Intervention
- Control Arm (No Intervention): Participants undergoing the control arm are presented with low-stress equivalents to the speech and mental arithmetic tasks from the experimental (high-stress) arm. For the speech task, participants are instructed to talk out loud to themselves for five minutes about a movie or book of their choice. Their speech is recorded using a small audio recorder device the research assistant prepares. For the mental arithmetic task, participants are instructed to count by increments of 15 starting from zero to the largest number they can reach. Participants are left in the room alone for the task for five minutes, after which the participant self-reports to the research assistant the number they reached.

INTERVENTIONS:
Behavioral: High-Stress Intervention — Those undergoing the High-Stress will be exposed to a gold-standard laboratory stressor, the Trier Social Stress Test (Kirschbaum et al., 1993), which reliably induces cortisol reactivity in most individuals.
  Arms: Experimental (High-Stress) Arm

SUMMARY:
This study will use a within-subjects design in a sample of individuals with a range of food insecurity recruited from the Los Angeles community (N = 400; 50% men). These participants will then, in counterbalanced order, be exposed to a gold-standard laboratory stressor and a control condition, one month apart. Moderation analyses will test whether cortisol reactivity to the stressor acts as a modulator of the relationship between high levels of food insecurity and increased hyperpalatable food intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* English-speaking

Exclusion Criteria:

* Recent (<1 year) diagnosis of major psychiatric disorders including any mood disorder, schizophrenia, or PTSD
* Recent (<1 year) diagnosis of eating disorder
* Recent (<1 year) diagnosis of metabolic or endocrine disorder or steroid or hormonal contraceptive use
* Pregnancy
* Allergy to any of the foods in the food buffet
* Participation in strict dieting or caloric restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Hyperpalatable Food Intake Measured in Kilocalories | Hyperpalatable food intake will be measured immediately after the intervention.
  The primary outcome will be hyperpalatable food intake, initially measured in grams and converted into kilocalories. The food will consist of the following items: donuts, M&Ms, potato chips, crackers, and Sprite. These foods were chosen because processed foods, added sugars, refined grains, starchy vegetables, and sugar sweetened beverages are foods to avoid according to the 2019 American Diabetes Association Nutrition Consensus Report and are high in carbohydrates and glycemic index.

CONTACTS AND LOCATIONS:
Overall Officials: A. Janet Tomiyama, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] American Diabetes Association. Diabetes care standards of medical care in Diabetes - 2019. J Clin Appl Res Educ 2019.